CLINICAL TRIAL: NCT05448573
Title: Müdigkeit Und Erschöpfung Rechtzeitig Erkennen Und LINdern - a Longitudinal Study to Investigate and Develop a Patient-centered and Effective Fatigue Screening
Brief Title: A Longitudinal Study to Investigate and Develop a Patient-centered and Effective Fatigue Screening
Acronym: MERLIN
Status: Active, not recruiting | Type: Observational
Sponsor: German Cancer Research Center (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Sponsor
Other Study IDs: MERLIN
Record Dates: First submitted 2022-06-13; First posted 2022-07-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Cancer-related Fatigue
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Fatigue Screening and assessment — (Newly) diagnosed cancer-patients from any cancer entity. No intervention.

SUMMARY:
MERLIN will include 300 cancer patients at the beginning of their systemic cancer therapy. Patients' fatigue-levels will be surveyed at short time intervals during their cancer therapy and at longer intervals during the subsequent post-treatment phase.

DETAILED DESCRIPTION:
MERLIN aims to answer the question, how a fatigue screening tool should be designed for use in clinical practice to reliably and efficiently detect fatigue in cancer patients.

Patients will be surveyed at short time intervals during their cancer therapy (every 1-2 weeks) and at longer intervals during the subsequent post-treatment phase (every 4-6 weeks).

In addition, important psychological factors, which may exacerbate fatigue or contribute to its maintenance will be assessed at baseline, after 3, 6, 12 and 18 months (e.g. depressive symptoms, anxiety, sleep disturbances, coping). These data will be collected by online questionnaires.

Additional data, e.g. medical history, cancer characteristics and treatment as well as concomitant medication and complementary therapies will be extracted from the clinical documentation systems.

In total, the study will provide important information for the establishment of a patient-oriented fatigue screening. Thus, MERLIN will contribute to the early detection and alleviation of this frequent and distressing side effect of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* having received a cancer diagnosis (any entity, any stage)
* before or within the first month of systemic therapy or radiotherapy against this cancer
* age ≥ 18 years
* having the ability to consent to the study

Exclusion Criteria:

* previous systemic cancer therapies or radiotherapy within the last 6 months
* diagnosis of chronic fatigue syndrome / myeloid encephalitis
* unable to understand the study protocol and complete scheduled assessments during the study period (e.g., for language, cognitive, medical, or organizational reasons)
* not able to complete the survey online via smartphone, PC, or tablet

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients from any cancer entity at any cancer stage
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
1st fatigue screening | Baseline - 18 months
  based on the first Cella-criterion, 3 (dichotomous) items
2nd fatigue screening | Baseline - 18 months
  Visual Analogue Scale (VAS) for Energy, 1 item (Numeric Rating Scale 0-10), higher values meaning higher energy levels.
3rd fatigue screening | Baseline - 18 months
  short Fatigue impact, 1 item (Numeric Rating Scale 0-10), higher values meaning higher fatigue impact on daily functioning.
Cancer-related fatigue (as reference criterion) | Baseline - 18 months
  based on Cella criteria, 11 (dichotomous) items

SECONDARY OUTCOMES:
Multidimensional fatigue | Baseline - 18 months
  EORTC QLQ - FA12 (physical, emotional, and cognitive dimension). The items are rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much) with higher scores meaning a higher level of fatigue.
Fatigue impact | Baseline - 18 months
  Brief Fatigue Inventory (BFI). The BFI consists of an 11-point numerical rating scale ranging from 0 (no fatigue) to 10 (as bad as you can imagine) with higher scores signifying higher intensity and impairment
Quality of life, function and symptoms | Baseline - 18 months
  assessed by the EORTC QLQ-C30. The items are rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much). A higher score corresponds to a higher level of symptoms/problems
Depressive symptoms and anxiety | Baseline - 18 months
  assessed by the Patient Health Questionnaire (PHQ-4), 4 items. The items are rated on a 4-point scale ranging from 0 (not at all) to 3 (most of the time). A sum score is calculated, with higher scores meaning a higher level of depressive symptoms and anxiety
Physical activity | Baseline - 18 months
  assessed by a questionnaire regarding walking, cycling, and exercise behavior
Sleep disorders | Baseline - 18 months
  assessed by the PSQI (Pittsburgh Sleep Quality Index).The PSQI consists of open and closed questions regarding characteristics of sleep and sleep quality. Some items are rated on a 4-point likert scale with higher scores meaning more sleep problems.
Fatigue Coping | 3 months - 18 months
  assessed by an adapted Brief COPE questionnaire. The questionnaire consists of 14 items and the items are rated on a 4-point Likert scale with higher scores meaning higher use of the coping strategy described
Distress | Baseline - 18 months
  assessed by the Distress Thermometer, 0-10 Numerous Rating scale. Higher values meaning more distress
Occupational Issues (Past) | T4 (18 months)
  Pre-diagnosis working status, 2 items
Occupational Issues (Present) | T4 (18 months)
  Current working status, 4 items
EORTC single item | Baseline - 18 months
  suffering from hot flashes, 4-point Likert scale. A higher value means more suffering.
Social Support | Baseline - 18 months
  assessed by the Illness-specific Social Support Scale (ISSS, German Version) among cancer patients. The 8 items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (always). Sum scores for the items 1,3,6 and 8 (positive support) as well as for the items 2,4,5 and 7 (detrimental interaction) are calculated with higher scores meaning higher levels of positive support and detrimental interaction respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Steindorf, Prof. Dr., Principal Investigator — German Cancer Research Center, C110, Heidelberg, Baden-Württemberg, Germany; Martina E. Schmidt, Dr., Principal Investigator — German Cancer Research Center, C110, Heidelberg, Baden-Württemberg, Germany; Alexander Haussmann, Dr., Principal Investigator — German Cancer Research Center, C110, Heidelberg, Baden-Württemberg, Germany; Anne Katrin Berger, Prof. Dr., Principal Investigator — National Center for Tumor Diseases (NCT), University Hospital Heidelberg, Heidelberg, Germany
Locations (1):
- German Cancer Research Center, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blickle P, Haussmann A, Holzner B, Berger AK, Steindorf K, Schmidt ME. Providing the basis for a patient-centred and effective screening for cancer-related fatigue (MERLIN study): design of a longitudinal observational study. BMJ Open. 2023 Sep 28;13(9):e073802. doi: 10.1136/bmjopen-2023-073802. PMID 37770278